CLINICAL TRIAL: NCT06918418
Title: Comparison of Salbutamol Alone and Salbutamol in Combination With Ipratropium Bromide in Treatment of Acute Asthma in Children
Brief Title: A Comparative Study of Adding Ipratropium to Salbutamol for the Treatment of Asthma Attack in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital and Institute of Child Health, Multan (Other Government)
Responsible Party: Principal Investigator, Muhammad Umair, Principal Investigator, Children's Hospital and Institute of Child Health, Multan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1321-1030
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Asthma Exacerbation; Children
Keywords: Asthma; Salbutamol; Ipratropium Bromide; Pulmonary Asthma Score
MeSH Terms: conditions — Asthma | interventions — Albuterol; Ipratropium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Nebulization (Experimental): Combined Salbutamol and Ipratropium Bromide
  Interventions: Drug: salbutamol + ipratropium bromide nebules
- Single Nebulization (Active Comparator): Salbutamol Nebulization alone
  Interventions: Drug: Salbutamol (Ventolin®)

INTERVENTIONS:
Drug: Salbutamol (Ventolin®) — Children were given 0.5% salbutamol aerosol solution (0.15 mg/kg weight, up to a maximum of 5 mg) in 5mL of normal saline solution for 7 min every 20 min for 2 h, and then every 30 min for two more hours. Aerosol were generated by nebulizer powered by compressed-air (5 L/min) with Y-connection with oxygen (3 L/min) and delivered via a face mask.
  Other Names: Albuterol
  Arms: Single Nebulization
Drug: salbutamol + ipratropium bromide nebules — In addition to Salbutamol nebulization, children received ipratropium bromide nebulization. Ipratropium bromide solution (250 mcg in children <20 kg weight or 500 mcg in children >=20 kg) every 20 min for the first 2 hours then every 30 min for 2 hours more will be given in between the salbutamol nebulization. Aerosol were generated by nebulizer powered by compressed-air (5 L/min) with Y-connection with oxygen (3 L/min) and delivered via a face mask.
  Other Names: Albuterol; Atrovent
  Arms: Combined Nebulization

SUMMARY:
The goal of this clinical trial was to determine if adding ipratropium bromide to salbutamol improves asthma treatment in children.

The main question this study aimed to answer was:

Does combining ipratropium with salbutamol improve asthma symptoms more effectively than salbutamol alone?

Researchers compared salbutamol alone to a combination of salbutamol and ipratropium in children with acute asthma.

Participants:

(i) Received either salbutamol alone or salbutamol with ipratropium via nebulization for 4 hours

(ii) Had their asthma symptoms assessed before and after treatment

(iii) Were discharged with continued treatment and counseling if stable

This study was conducted in the Department of Pediatric Medicine, Children's Hospital Multan, over six months. A total of 60 children with acute asthma were included.

DETAILED DESCRIPTION:
Children presenting with asthma exacerbation were assessed for eligibility. Eligible participants had their baseline characteristics recorded including age, gender, history of parental asthma, duration of asthma diagnosis, use of asthma controllers (inhaled corticosteroids, Long Acting Beta Agonist (LABA), Montelukast) & baseline pulmonary asthma score. Through lottery method using sequentially numbered sealed opaque envelopes children were assigned to group A and group B treatments. At the end of 4-hours of therapy, pulmonary asthma score was re-assessed by pediatrician not aware of treatment assigned. Once stabilized, the children were discharged on regular nebulization therapy with controller medication after proper counseling.

ELIGIBILITY:
Inclusion Criteria:

* Children with acute asthma exacerbation (presenting with wheeze, labored breathing with ronchi audible on auscultation)
* Within 12 hours of symptom onset

Exclusion Criteria:

* Children with known pulmonary and/or cardiac congenital malformations
* Bronchopulmonary dysplasia
* Cystic fibrosis
* Post infectious bronchiolitis obliterans
* Altered mental status on presentation with imminent respiratory failure (pulmonary asthma score ≥ 10, cases needing PICU care)

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Pulmonary Asthma Score (PAS) | On presentation and four hours after treatment.
  Asthma severity was assessed using Pulmonary Asthma score. It uses respiratory rate, wheezing, inspiration to expiration ratio (I:E) and use of accessory muscles graded 0 - 3 with total score of 12.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Muhammad Aslam Sheikh, FCPS, Study Chair — Children's Hospital and Institute of Child Health, Multan
Locations (1):
- Children's Hospital and Institute of Child Health, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Since the study involves children, there are strict ethical guidelines regarding data privacy and protection of minors' health information. Sharing detailed IPD may risk re-identification.

REFERENCES:
- [Background] Iramain R, Lopez-Herce J, Coronel J, Spitters C, Guggiari J, Bogado N. Inhaled salbutamol plus ipratropium in moderate and severe asthma crises in children. J Asthma. 2011 Apr;48(3):298-303. doi: 10.3109/02770903.2011.555037. Epub 2011 Feb 21. PMID 21332430
- [Background] Memon BN, Parkash A, Ahmed Khan KM, Gowa MA, Bai C. Response to nebulized salbutamol versus combination with ipratropium bromide in children with acute severe asthma. J Pak Med Assoc. 2016 Mar;66(3):243-6. PMID 26968269